CLINICAL TRIAL: NCT03533205
Title: Prediction of Hemodynamic Instability in Patients Undergoing Surgery
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, D.P.Veelo, MD PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: W15_080
Record Dates: First submitted 2018-04-26; First posted 2018-05-23 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Blood Pressure; Prediction Models; Machine Learning; Hemodynamic Instability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Hypotension Probability Indicator — The accurary of the Hypotension Probability Indicator (HPI) is tested in the created offline database. This means data was prospectively collected but the HPI algorithm was not tested prospectively but after collection in the offline database.

SUMMARY:
Intraoperative hypotension occurs often and is associated with adverse patient outcomes such as stroke, myocardial infarction and renal injury.

The aim of this study was to test the accuracy of a physiology-based machine-learning algorithm using continuous non-invasive measurement of the blood pressure waveform with the Nexfin® finger cuff during surgery.

ELIGIBILITY:
Inclusion Criteria:

* all adult patients undergoing surgery

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adult patients undergoing surgery in the AMC were included in the study. Subjects were only excluded when technical problems or strong local vasoconstriction (i.e., cold fingers) prevented the Nexfin® non-invasive blood pressure finger cuff measurement. Subjects were not excluded for any other reason besides technical failure.
Sampling Method: Non-Probability Sample
Enrollment: 507 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2018-04-26 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the HPI algorithm | three minutes prior to the hypotensive event
  Sensitivity
Specifity of the HPI algorithm | three minutes prior to the hypotensive event
  Specifity

SECONDARY OUTCOMES:
Predictive positive value of the HPI algorithm | one minute prior to the hypotensive event
  Predictive positive value
Predictive positive value of the HPI algorithm | two minutes prior to the hypotensive event
  Predictive positive value
Predictive positive value of the HPI algorithm | three minutes prior to the hypotensive event
  Predictive positive value
Predictive positive value of the HPI algorithm | four minutes prior to the hypotensive event
  Predictive positive value
Predictive positive value of the HPI algorithm | five minutes prior to the hypotensive event
  Predictive positive value
Predictive positive value of the HPI algorithm | ten minutes prior to the hypotensive event
  Predictive positive value
Predictive positive value of the HPI algorithm | 15 minutes prior to the hypotensive event
  Predictive positive value
Negative predictive value of the HPI algorithm | one minute prior to the hypotensive event
  Negative predictive value
Negative predictive value of the HPI algorithm | two minutes prior to the hypotensive event
  Negative predictive value
Negative predictive value of the HPI algorithm | four minutes prior to the hypotensive event
  Negative predictive value
Negative predictive value of the HPI algorithm | five minutes prior to the hypotensive event
  Negative predictive value
Negative predictive value of the HPI algorithm | ten minutes prior to the hypotensive event
  Negative predictive value
Negative predictive value of the HPI algorithm | 15 minutes prior to the hypotensive event
  Negative predictive value
Time from HPI alarm to hypotensive event during surgery | From the onset of the HPI alarm to the hypotensive event during surgery, this is in minutes. (this can range from 0,1 min to a high number such as 30 or even 40 minutes)
  Time from HPI alarm to hypotensive event, this can range from 0,1 min to a high number such as 30 or even 40 minutes.
Sensitivity of the HPI algorithm | one minute prior to the hypotensive event
  Sensitivity
Sensitivity of the HPI algorithm | two minutes prior to the hypotensive event
  Sensitivity
Sensitivity of the HPI algorithm | five minutes prior to the hypotensive event
  Sensitivity
Sensitivity of the HPI algorithm | ten minutes prior to the hypotensive event
  Sensitivity
Sensitivity of the HPI algorithm | 15 minutes prior to the hypotensive event
  Sensitivity
Specifity of the HPI algorithm | one minute prior to the hypotensive event
  Specifity
Specifity of the HPI algorithm | two minutes prior to the hypotensive event
  Specifity
Specifity of the HPI algorithm | five minutes prior to the hypotensive event
  Specifity
Specifity of the HPI algorithm | ten minutes prior to the hypotensive event
  Specifity
Specifity of the HPI algorithm | 15 minutes prior to the hypotensive event
  Specifity

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wijnberge M, van der Ster BJP, Geerts BF, de Beer F, Beurskens C, Emal D, Hollmann MW, Vlaar APJ, Veelo DP. Clinical performance of a machine-learning algorithm to predict intra-operative hypotension with noninvasive arterial pressure waveforms: A cohort study. Eur J Anaesthesiol. 2021 Jun 1;38(6):609-615. doi: 10.1097/EJA.0000000000001521. PMID 33927105